CLINICAL TRIAL: NCT01339520
Title: Use of a Card to Improve Risk Factor Control in Patients With Type II Diabetes
Brief Title: Diabetes Scorecard Educational Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Michael Irwig, Attending Physician, George Washington University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DiabetesScorecardStudy
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scorecard (Experimental): Score of points for variables.
  Interventions: Behavioral: Scorecard; Behavioral: Control
- Control (No Intervention): Standard of care for diabetes subjects

INTERVENTIONS:
Behavioral: Scorecard — Points were assigned for blood pressure, HbA1c level, LDL-cholesterol level, aspirin use and exercise level.
  Arms: Scorecard
Behavioral: Control — Standard of care for diabetes subjects
  Arms: Scorecard

SUMMARY:
The purpose of this study is to see if the use of a diabetic scorecard during clinic visits can improve glycemic control, blood pressure control, LDL-cholesterol, aspirin usage, and amount of exercise in adults over age 40 with uncontrolled Type II diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled Type II diabetes (HbA1c ≥ 8%)

Exclusion Criteria:

* Type I Diabetes
* HbA1c < 8%
* Inability to understand the diabetes scorecard due to condition (i.e. dementia, mental retardation, etc) or language barrier
* Pregnancy
* Planning to move within the next year

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in total score | 9 months
  The total score was calculated by points assigned to variables (systolic blood pressure, diastolic blood pressure, HbA1c, aspirin usage and daily exercise). The maximal score of 100 corresponds to all variables at target. Fewer points were assigned to higher blood pressure, worse HbA1c levels, less exercise, etc.

SECONDARY OUTCOMES:
LDL-cholesterol | 9 months
HbA1c | 9 months
  Measure of glycemic control

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty Associates, George Washington University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Irwig MS, Sood P, Ni D, Amass T, Khurana PS, Jayanthi VV, Wang L, Adler SM. A diabetes scorecard does not improve HbA(1c), blood pressure, lipids, aspirin usage, exercise and diabetes knowledge over 9 months: a randomized controlled trial. Diabet Med. 2012 Sep;29(9):1206-12. doi: 10.1111/j.1464-5491.2012.03610.x. PMID 22332914